CLINICAL TRIAL: NCT07013136
Title: Efficacy and Safety of Folic Acid on Acute Kidney Injury in Adults: A Feasibility Study
Brief Title: Feasibility Test of Folic Acid on Acute Kidney Injury
Acronym: Folate_AKI
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Folate_AKI-RAINER-2024
Record Dates: First submitted 2025-04-25; First posted 2025-06-10 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-04

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Clinical trial; Feasibility study; Folate; 5-Methyltetrahydrofolate; Repurpose
MeSH Terms: conditions — Acute Kidney Injury | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1. Usual care (No Intervention): Usual care is given until AKI is resolved.
- Arm 2. Folic acid 5 mg + Usual care (Experimental): Oral folic acid 5mg is given once a day until AKI is resolved*, to a maximum of 30 days**.
  Interventions: Drug: Folic Acid 5 MG

INTERVENTIONS:
Drug: Folic Acid 5 MG — In this study, oral folic acid at 5 mg/d (~83.3 μg/kg) is chosen. In a rat model of AKI with ischaemia-reperfusion, intraperitoneal injection of 5-methyltetrahydrofolate (5-MTHF) at 3 μg/kg body weight twice (30 min before ischaemia and 3 h after reperfusion) improved kidney function and alleviated oxidative stress within 24 hours. The average body weight is around 60 kg for Chinese. Considering the oral route often requires larger doses than injection to produce the same effect, oral folic acid at 5 mg/d (~83.3 μg/kg) is chosen to test its effect on AKI. Depending on the clinical condition, the therapeutic dose of folic acid varies. For foetal support during pregnancy, daily doses of 1 mg of folic acid are recommended; for lowering homocysteine, up to 5 mg daily are generally used.
  Arms: Arm 2. Folic acid 5 mg + Usual care

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility of folic acid supplementation as a treatment for adult patients with acute kidney injury (AKI) receiving hospital care.

The main question it aims to answer is: Is it feasible to conduct a fully-powered randomized controlled trial (RCT) to assess the efficacy and safety of folic acid supplementation in AKI management?

Researchers will compare two groups (usual care vs. usual care + 5 mg folic acid) to determine the feasibility of folic acid supplementation and estimate the sample size required for a fully powered RCT.

Participants will:

1. Receive either usual care, or usual care combined with oral folic acid (5 mg daily) until AKI resolution (up to 30 days);
2. Undergo regular monitoring during hospitalization and follow-ups at 3 months and one year post-discharge.

DETAILED DESCRIPTION:
1. Background Information

   Acute Kidney Injury (AKI) is a worldwide health issue affecting over 13 million people each year with a significant hospital mortality of 20-40%. It is characterized by an abrupt loss of kidney function and is associated with multiple long-term sequelae including chronic kidney disease (CKD) and reliance on renal replacement therapy (RRT). Patients with AKI place a substantial financial burden on healthcare resources. In England, the annual cost of AKI is estimated at £1 billion, consuming 1% of the National Health Service (NHS) budget; in the United States (US), inpatient AKI costs $5 to $24 billion per year. However, there are few therapies to moderate the risk and long-term sequelae of AKI. Timely, efficient treatment of AKI will benefit both patients and health care systems.

   The National Confidential Enquiry into Patient Outcome and Death (NCEPOD) report on hospital mortality primarily due to AKI judges that good clinical practice occurred in only 50% cases, 33% patients were under insufficient investigations, 29% patients received inadequate clinical management, and complications were badly handled in over 50% cases. Progression of the admission stage of AKI to a higher stage was reported to be associated with a 39% inpatient mortality compared with a 21% mortality in those who did not progress. If the AKI stage could be prevented to deteriorate to a higher stage, the mortality rate of AKI patients during hospital stay would drop almost half.

   1.1 Epidemiology, Etiology and Pathophysiology of AKI AKI is a common problem in all countries of the world, and its prevalence has been reported to range from <1% to 66%. Apart from population differences, different classification systems used in epidemiological studies also conduced to the varied estimation of AKI incidence. Little epidemiological data is available for AKI in Hong Kong (HK). Szeto reported a crude hospital admission of AKI of 12% amongst 140,000 hospital admissions observed in a tertiary referral center of HK. The crude mortality rate of AKI in patients attending an emergency department (ED) in HK is 25%.

   AKI is a multifactorial syndrome. The causes of AKI can be classified into three categories: prerenal, intrinsic renal and postrenal. Prerenal causes involve reduced renal perfusion due to medication, sepsis or volume depletion (e.g., diuretic overuse and diarrhea). Intrinsic renal causes typically result from infections, prolonged hypotension, nephrotoxic drugs or pre-existing renal impairment (e.g., glomerulonephritis and vasculitis). Postrenal AKI is due to obstruction of urinary flow, especially common in elderly men. Sepsis, infection and use of nephrotoxic drugs are common causes of AKI overall, leading to reduced renal blood flow. Sepsis is the most common contributor to AKI (25%). In intensive care unit (ICU) settings, AKI was found to occur in more than half of patients, and half of all patients with AKI in ICU have sepsis. Drug induced AKI occurs in 20% of hospital cases, and those drugs include non-steroidal anti-inflammatory drugs (NSAIDs), metformin, aminoglycosides, angiotensin converting enzyme inhibitors (ACEI), angiotensin II receptor blockers (ARBs), diuretics and iodine containing X-ray contrast. In low-to-middle-income settings, environmental factors such as endemic infections (e.g., malaria and dengue fever) and contaminated water are also common factors to induce AKI.

   The diverse etiologies of AKI along with other comorbidities make it difficult to determine and understand the pathophysiology of AKI. Recently, oxidative stress has been accepted as the primary mediator of adverse outcomes in AKI, playing a critical role in both initiating and further development of AKI. In the context of deficient renal blood flow in AKI, ischemia-reperfusion represents the most common mechanism in which oxygen and nutrient delivery as well as waste removal are impaired; this mismatch of oxygen supply and demand, and accumulation of waste lead to cellular injury and even death. Sepsis-induced AKI also triggers oxidative stress. Oxidative stress as a key component in the pathophysiology of AKI provides a target for potential therapeutics.

   Currently, the KDIGO serum creatinine-based criteria is mostly used to stage AKI. The KDIGO defines AKI as either an increase in serum creatinine to ≥1.5 times baseline or ≥0.3 mg/dl (≥26.5 μmol/l) within 48 hours. Depending on the cause and severity of AKI, the clinical presentation of patients with AKI varies. Mild to moderate AKI could be asymptomatic, and severe AKI could present clinical symptoms of uremia. AKI is a rapid (within 48 hours) loss of kidney function, and delays in detection and treatment may contribute to an in-hospital mortality rate of 20-40% that is higher than acute stroke and acute myocardial infarction combined.

   1.2 Treatment for AKI Management of AKI is primarily supportive, lacking effective therapeutic drugs. The key to management is assuring hemodynamic stability and preventing hypovolemia in patients so as to ensure sufficient renal perfusion. Depending on the cause and severity of AKI, treatments in hospital usually include: blood pressure and circulating electrolyte control; body fluid balance (e.g., with fluid replacement and/or diuretics); review and cessation of nephrotoxic medication; removing the obstruction if there's a blockage; and use of antibiotics. In severe cases, dialysis may be needed but dialysis is not disease-modifying. Malnutrition is a frequent problem in patients with AKI. Patients should follow a kidney-friendly eating plan to help the kidneys heal, maintain adequate nutrition and restrict potassium. There are no approved pharmacological agents for treating AKI.

   1.3 Folate Folic acid is a common external supplement of folate (Vitamin B9). Folic acid is a synthetic, parent compound of folate family. Folic acid gets metabolized into 5-methyltetrahydrofolate (5-MTHF). 5-MTHF is the biologically active form of folate and the predominant form of dietary folate in plasma.

   A systematic review was conducted in accordance with the PRISMA guidelines and registered in PROSPERO (CRD42024589377). The investigators searched six databases (PubMed, MEDLINE, CINAHL, CENTRAL, Embase, and Web of Science) from their inception until March 2024, identifying 36 randomized controlled trials (RCTs) that evaluated folate use in patients with CKD or AKI. Of these, 22 RCTs compared folate use with no use in patients with CKD, with treatment durations ranging from 4 weeks to 4.5 median years, and majority use folic acid. Notably, no published data focused on AKI populations. Among included RCTs, 20 reported that folate use significantly reduced homocysteine (Hcy) levels but not directly reduced cardiovascular events in CKD patients. Only 5 trials assessed markers of kidney disease progression including 3 measured serum creatinine and 2 measured estimated glomerular filtration rate (eGFR) with inconsistent findings. The largest study, China Stroke Primary Prevention Trial with 1671 CKD patients, demonstrated that folate use slowed the annual decline in eGFR compared to controls (0.96 ± 5.81% vs. 1.72 ± 6.08%, respectively). Similarly, a modest reduction in serum creatinine was observed in end-stage renal disease (ESRD) patients receiving folate (10.94 ± 2.01 vs. 11.30 ± 2.31 in controls). Safety analyses across all 22 RCTs revealed no severe adverse events attributable to folate, and no significant differences in adverse outcomes were noted between the treatment and control groups.

   Low doses: In a rat model of AKI with ischemia-reperfusion, 5-MTHF at a low dose of 3 μg/kg body weight improved kidney function, reduced plasma creatinine levels and alleviate oxidative stress within 24 hours. The expression of neutrophil gelatinase-associated lipocalin (NGAL), a marker of proximal tubular injury, was significantly reduced after folate treatment. 5-MTHF activated the nuclear factor erythroid 2-related factor 2 (Nrf2), a key regulator of the antioxidant defense system. Nrf2 activation regulates gene expression of detoxification enzymes and antioxidant proteins, which is vital to restore antioxidant defense against oxidative stress injury. Oxidative stress is the mainstay responsible to the adverse outcomes in AKI. The expression of antioxidant enzymes, superoxide dismutase-1 (SOD-1), glutathione synthesizing enzymes and heme oxygenase-1 (HO-1), were all upregulated after folate treatment.

   High doses: Folic acid, a precursor of folate, at high doses, e.g., 250 mg/ /kg body weight, has been used to induce AKI in animals. Folic acid causes AKI due to the rapid onset of folic acid crystals within renal tubules with a subsequent acute tubular necrosis, epithelial regeneration and renal cortical scarring. High concentrations of folic acid will lead to oxidative stress, mitochondrial abnormalities, ferroptosis, pyroptosis and increased expression of fibroblast growth factor 23 (FGF23). However, folic acid induced AKI is only experimental in animals, and high levels of folic acid have not been observed in the clinic kidney diseases.

   1.4 Unmet Clinical Need AKI is a common health issue with high morbidity and mortality in hospital. Delays in detection and treatment result in an in-hospital mortality rate of 20-40% that is higher than acute stroke and acute myocardial infarction combined. Management of AKI is primarily supportive. There are no approved pharmacological agents for treating AKI. Oxidative stress provides a target for therapeutics. Animal experiments have shown folate IN LOW DOSES alleviated oxidative stress, decreased plasma creatinine levels and improved kidney function of AKI. Folate administration has been studied to improve survival of patients with CKD using randomized clinical trials. Evidence for the protective effect of folate against AKI to safely reduce circulating creatinine levels, progression to CKD/ESRD and mortality in adult patients with AKI is needed.

   1.5 Impact If folate treatment improved outcome for 1% cases, as the global burden of AKI per year is 13 million cases, then potentially 130,000 patients could benefit per year; in HK, as AKI identiﬁed with a crude hospital admission of 12%, among around 2 million hospital admissions in one year, potentially 2,500 patients could benefit per year.
2. Aims and Hypotheses

   2.1 Aims This study aims to evaluate the folate intervention feasibility in adult patients with AKI, and the possibility of conducting a future fully powered RCT. The investigators propose to conduct this feasibility study among adults with AKI receiving usual care in the ED, ICU and medical wards at Queen Mary Hospital (QMH).

   2.2 Hypotheses The hypotheses of this study are set as meeting the feasibility criteria: ≥70% of patients recognized as eligible by clinicians are randomly allocated to study arm of which ≥70% of patients complete 90% or greater of the course of treatment and less than 5% adverse events (AEs) difference between no supplement control and folate supplement arms.
3. Plan of Investigation

This is a feasibility study with an open-label, randomized, 1:1 ratio (Usual care vs. 5 mg folic acid + Usual care).

This study will be conducted in accordance with Good Clinical Practice (GCP) guidelines and reported in accordance with the Consolidated Standards of Reporting Trials (CONSORT) statement.

3.1 Screening, recruitment and consent The investigators will check hospital records and the Clinical Management System (CMS) to identify potential participants. Then, the investigators will use a screening form to determine the eligibility of potential participants, and review their medical records. Eligible patients will be informed the study and asked for the consent to participate.

3.2 Randomization An investigator with no clinical involvement in the trial will do block randomization. The two study arms of control, and 5 mg/d folate will be allocated according to the randomization orders.

The study information and medications will be put into sealed envelopes. The outside of the envelope will contain the name of the study and possible arms contained within, but not which arm is selected. Each enrolled patient will be assigned an order number and receive the corresponding envelope. The patient ID, date, time and other information will be recorded on the envelope. Once the patients completed all baseline assessments, they will be allocated the treatment. In the case of broken or lost envelopes, the researcher figures out what the number of the envelope it is and replaces the envelope with the same treatment according to the allocation.

Hospital clinicians are responsible for administration of the allocated treatment. The patient's own doctors are free to modify or stop study treatment if they feel that it is in the best interests of the patient without the need for the patient to withdraw from the study.

3.3 Data collection An admission log, blood tests, investigations, medication review, and adverse events will be recorded for every patient. Screening form and consent form will be recorded for every patient. A member of the hospital clinical or research staff (as appropriate/designated) will collect this information and enter it into an IT system. The investigators will collect patient information before randomization and follow up daily for up to 30 days. Additional follow-ups will be conducted at 3 months and one year by contacting patients on the ward, in an outpatient setting, by phone or via their electronic record. Personal information and study data will be kept for 3 years after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for the study if ALL the following are present:

1. Adults ≥18 years of age;
2. AKI;
3. Intended or existing hospitalisation;
4. No medical history that might, in the opinion of the attending clinician, put the patient at significant risk if he/she were to participate in the study;
5. Informed consent

Exclusion Criteria:

Patients will be excluded from the study if any of the following conditions is present:

1. Refusal of consent expressed by the patient, close relative or legally appointed representative;
2. Enrolled in other research studies within previous 30 days;
3. Not expected to survive 3 days due to renal disease or other co-existing diseases;
4. Planned inter-hospital transfer within 3 days;
5. Recent surgery (<30 days);
6. Pregnancy;
7. Cardiac arrest prior to inclusion;
8. Contraindication to folate;
9. Already on folate treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of intervention | From enrollment to the end of treatment up to 30 days
  A preset feasibility goal of 70% or greater of recognized patients joining the study with 70% or more adherence to scheduled dosages of the intervention until AKI is resolved or to a maximum of 30 days [Binary Y/N].
30-day Severe Adverse Events | From enrollment to the end of treatment up to 30 days
  The incidence of severe adverse events (SAEs) in patients receiving folate supplementation [Binary Y/N].

SECONDARY OUTCOMES:
Screening rate | At enrollment
  Proportion of potential participants being screened for eligibility [Binary Y/N].
Consent rate | At enrollment
  Proportion of eligible participants signing the consent form to join the study [Binary Y/N].
Time from presentation to consent | At enrollment
  Time how long it takes to enroll a eligible participant from presentation to signing the consent form [Numerical].
Acceptability of a future randomized controlled trial (RCT) | From enrollment to the end of treatment up to 30 days
  The degree to which attending clinicians and patients are willing to participate in a fully-powered RCT in the future [Numerical Score: 0 - 10, higher scores mean a better outcome].
Retrieval rate of patient outcomes | From enrollment to the end of treatment at 30 days, 3 months and one year
  The percentage of patients successfully followed up for outcome reporting [Binary Y/N].
AKI recovery | From enrollment to the end of treatment up to 30 days
  Proportion of recovery versus progression to a severer stage of AKI or AKD in each treatment arm [Binary Y/N].
Duration of hospitalization | From enrollment to the end of treatment up to 30 days
  Total length of time a patient remains admitted to a hospital [Numerical].
Need of renal replacement therapy (RRT) | From enrollment to the end of treatment up to 30 days
  Proportion of patients requiring RRT to support kidney function in each treatment arm [Binary Y/N].
Kidney function at 3 months post-AKI | At 3 months
  The recovery status of renal function following treatment at 3 months (classified as full recovery, partial recovery, persistent impairment, and progression to CKD).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H Rainer, MBBCh, Principal Investigator — Department of Emergency Medicine, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shelton LM, Park BK, Copple IM. Role of Nrf2 in protection against acute kidney injury. Kidney Int. 2013 Dec;84(6):1090-5. doi: 10.1038/ki.2013.248. Epub 2013 Jun 19. PMID 23783243
- [Background] Pietrzik K, Bailey L, Shane B. Folic acid and L-5-methyltetrahydrofolate: comparison of clinical pharmacokinetics and pharmacodynamics. Clin Pharmacokinet. 2010 Aug;49(8):535-48. doi: 10.2165/11532990-000000000-00000. PMID 20608755
- [Background] Scaglione F, Panzavolta G. Folate, folic acid and 5-methyltetrahydrofolate are not the same thing. Xenobiotica. 2014 May;44(5):480-8. doi: 10.3109/00498254.2013.845705. Epub 2014 Feb 4. PMID 24494987
- [Background] Nikolic T, Petrovic D, Matic S, Turnic TN, Jeremic J, Radonjic K, Srejovic I, Zivkovic V, Bolevich S, Bolevich S, Jakovljevic V. The influence of folic acid-induced acute kidney injury on cardiac function and redox status in rats. Naunyn Schmiedebergs Arch Pharmacol. 2020 Jan;393(1):99-109. doi: 10.1007/s00210-019-01717-z. Epub 2019 Aug 27. PMID 31455992
- [Background] Matsuura R, Doi K, Rabb H. Acute kidney injury and distant organ dysfunction-network system analysis. Kidney Int. 2023 Jun;103(6):1041-1055. doi: 10.1016/j.kint.2023.03.025. Epub 2023 Apr 6. PMID 37030663
- [Background] Thomas ME, Blaine C, Dawnay A, Devonald MA, Ftouh S, Laing C, Latchem S, Lewington A, Milford DV, Ostermann M. The definition of acute kidney injury and its use in practice. Kidney Int. 2015 Jan;87(1):62-73. doi: 10.1038/ki.2014.328. Epub 2014 Oct 15. PMID 25317932
- [Background] Yan LJ. Folic acid-induced animal model of kidney disease. Animal Model Exp Med. 2021 Nov 24;4(4):329-342. doi: 10.1002/ame2.12194. eCollection 2021 Dec. PMID 34977484
- [Background] Sharfuddin AA, Molitoris BA. Pathophysiology of ischemic acute kidney injury. Nat Rev Nephrol. 2011 Apr;7(4):189-200. doi: 10.1038/nrneph.2011.16. Epub 2011 Mar 1. PMID 21364518
- [Background] Rahman M, Shad F, Smith MC. Acute kidney injury: a guide to diagnosis and management. Am Fam Physician. 2012 Oct 1;86(7):631-9. PMID 23062091
- [Background] Szeto CC. Perspectives on acute kidney injury strategy: Hong Kong. Nephrology (Carlton). 2018 Oct;23 Suppl 4:104-106. doi: 10.1111/nep.13450. PMID 30298652
- [Background] Hoste EAJ, Kellum JA, Selby NM, Zarbock A, Palevsky PM, Bagshaw SM, Goldstein SL, Cerda J, Chawla LS. Global epidemiology and outcomes of acute kidney injury. Nat Rev Nephrol. 2018 Oct;14(10):607-625. doi: 10.1038/s41581-018-0052-0. PMID 30135570
- [Background] Dasta JF, Kane-Gill S. Review of the Literature on the Costs Associated With Acute Kidney Injury. J Pharm Pract. 2019 Jun;32(3):292-302. doi: 10.1177/0897190019852556. PMID 31291842
- [Background] Negi S, Koreeda D, Kobayashi S, Yano T, Tatsuta K, Mima T, Shigematsu T, Ohya M. Acute kidney injury: Epidemiology, outcomes, complications, and therapeutic strategies. Semin Dial. 2018 Sep;31(5):519-527. doi: 10.1111/sdi.12705. Epub 2018 May 8. PMID 29738093
- [Background] Lameire NH, Bagga A, Cruz D, De Maeseneer J, Endre Z, Kellum JA, Liu KD, Mehta RL, Pannu N, Van Biesen W, Vanholder R. Acute kidney injury: an increasing global concern. Lancet. 2013 Jul 13;382(9887):170-9. doi: 10.1016/S0140-6736(13)60647-9. Epub 2013 May 31. PMID 23727171